CLINICAL TRIAL: NCT04072627
Title: Evaluation of Microbial Composition in Human Milk From Healthy Women in the Turkish Population: an Observational Cross-sectional Study
Brief Title: Microbial Composition of Breast Milk Collected From Healthy Turkish Women
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Collaborators: Turkish Society of Clinical Enteral and Parenteral Nutrition (Other)
Responsible Party: Principal Investigator, F. Gülhan Samur, Prof. Dr., Hacettepe University
Other Study IDs: Hacettepe Nutrition Diet
Record Dates: First submitted 2019-08-27; First posted 2019-08-28 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Microbial Community in Breast Milk
Keywords: breast milk; microbiota

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Breast Milk
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Breast milk is an optimal source of nutrients for newborns as well as a potential source of bacteria for the intestinal microbiota. However, there are limited number of studies evaluating the relationship between maternal nutrition, breast milk and neonatal intestinal microbiota.

DETAILED DESCRIPTION:
The study was conducted on a total of 20 healthy women following at Obstetrics and Gynecology Department of Gülhane Education and Research Hospital in Ankara Health Sciences University. Sociodemographic characteristics, anthropometric measurements, breastfeeding characteristics were evaluated in the third trimester of the women who underwent routine prenatal care. Breast milk samples were obtained at 16.day postpartum during lactation.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy
* Age 19-35 years
* At weeks of 30-36 gestation
* No history of acute or chronic diseases
* Term delivery

Exclusion Criteria:

* Alcohol use
* Smoking
* Gestational diabetes
* Type 1 and 2 diabetes
* Preeclampsia
* Polycystic ovary
* Syndrome
* Thyroid and parathyroid disease
* Metabolic bone or kidney disease
* Abnormal liver function
* Multiple pregnancy
* Premature and postmature labor
* Having chemotherapy
* Taking drugs such as antibiotics and probiotics

Ages: 20 Years to 31 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 20 healthy women who were at 16. day postpartum
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2018-05-05 (Actual); Primary Completion 2018-09-05 (Actual); Study Completion 2019-07-05 (Actual)

PRIMARY OUTCOMES:
Microbial abundance and diversity | at 16 day postpartum
  The microbial composition of the breast milk samples was determined by 16S rRNA (ribosomal ribonucleic acid) gene sequencing analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Gülhan SAMUR, Professor, Principal Investigator — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Murphy K, Curley D, O'Callaghan TF, O'Shea CA, Dempsey EM, O'Toole PW, Ross RP, Ryan CA, Stanton C. The Composition of Human Milk and Infant Faecal Microbiota Over the First Three Months of Life: A Pilot Study. Sci Rep. 2017 Jan 17;7:40597. doi: 10.1038/srep40597. PMID 28094284
- [Result] Fitzstevens JL, Smith KC, Hagadorn JI, Caimano MJ, Matson AP, Brownell EA. Systematic Review of the Human Milk Microbiota. Nutr Clin Pract. 2017 Jun;32(3):354-364. doi: 10.1177/0884533616670150. Epub 2016 Sep 27. PMID 27679525
- [Result] Jost T, Lacroix C, Braegger C, Chassard C. Assessment of bacterial diversity in breast milk using culture-dependent and culture-independent approaches. Br J Nutr. 2013 Oct;110(7):1253-62. doi: 10.1017/S0007114513000597. Epub 2013 Mar 14. PMID 23507238
- [Result] Hunt KM, Foster JA, Forney LJ, Schutte UM, Beck DL, Abdo Z, Fox LK, Williams JE, McGuire MK, McGuire MA. Characterization of the diversity and temporal stability of bacterial communities in human milk. PLoS One. 2011;6(6):e21313. doi: 10.1371/journal.pone.0021313. Epub 2011 Jun 17. PMID 21695057
- [Result] Chen PW, Lin YL, Huang MS. Profiles of commensal and opportunistic bacteria in human milk from healthy donors in Taiwan. J Food Drug Anal. 2018 Oct;26(4):1235-1244. doi: 10.1016/j.jfda.2018.03.004. Epub 2018 Apr 5. PMID 30249322
- [Result] Damaceno QS, Souza JP, Nicoli JR, Paula RL, Assis GB, Figueiredo HC, Azevedo V, Martins FS. Evaluation of Potential Probiotics Isolated from Human Milk and Colostrum. Probiotics Antimicrob Proteins. 2017 Dec;9(4):371-379. doi: 10.1007/s12602-017-9270-1. PMID 28374172